CLINICAL TRIAL: NCT04433195
Title: Xpert MTB/RIF Test as the Initial Diagnostic Test in the Diagnosis of Pulmonary Tuberculosis: a Pragmatic Trial
Brief Title: Xpert MTB/RIF Test in the Diagnosis of Pulmonary Tuberculosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Buddhist Tzu Chi General Hospital (Other); Chest Hospital, Ministry of Health and Welfare, Taiwan (Other Government); Chang-Hua Hospital (Other Government); Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: N202002038
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Tuberculosis Confirmation by Culture
Keywords: Tuberculosis; Xpert MTB/RIF; diagnostic turnaround time
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: pragmatic trial
Masking Description: both care providers and participants will be informed of positive results of Xpert MTB/RIF test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Immediate NAA by clinician (Active Comparator): Nucleic acid amplification test requested by clinicians as the initial diagnostic test for the diagnosis of pulmonary TB
  Interventions: Diagnostic Test: Xpert MTB/RIF test
- Immediate NAA as intervention (Experimental): Nucleic acid amplification test not requested by clinicians as the initial diagnostic test for the diagnosis of pulmonary TB, but Xpert MTB/RIF is performed as intervention in this study (intervention group)
  Interventions: Diagnostic Test: Xpert MTB/RIF test
- No immediate NAA (No Intervention): Nucleic acid amplification test not requested by clinicians as the initial diagnostic test for the diagnosis of pulmonary TB, and Xpert MTB/RIF is not performed as the initial diagnostic test in this study (control group). Nucleic acid amplification test may be ordered at a later point in time by clinicians as an add-on test after sputum smear microscopy

INTERVENTIONS:
Diagnostic Test: Xpert MTB/RIF test — Xpert MTB/RIF performed as the initial diagnostic test for the diagnosis of pulmonary TB
  Other Names: nucleic acid amplification test
  Arms: Immediate NAA as intervention; Immediate NAA by clinician

SUMMARY:
Currently in Taiwan, most clinicians use sputum smear and culture for the diagnosis of pulmonary tuberculosis (TB) and apply nucleic acid amplification (NAA) test in a selected manner. In 2013, the World Health Organization issued conditional recommendation that Xpert MTB/RIF may be used rather than conventional microscopy and culture as the initial diagnostic test in all adults suspected of having TB. The newly published Taiwan guidelines for TB diagnosis and treatment has recommended NAA test, together with smear and culture, as the initial diagnostic test in individuals suspected of having TB. The investigators conduct a prospective study to investigate the use of Xpert MTB/RIF as the initial diagnostic test of pulmonary TB under a pragmatic trial design.

DETAILED DESCRIPTION:
In this study the investigators will respect current practice in the use of NAA in the diagnosis of pulmonary TB. Clinicians may have ordered NAA as the initial diagnostic test in adults suspected of having pulmonary TB (group A, Immediate NAA by clinician), and the investigators will not intervene. For patients who do not have NAA as the initial diagnostic test, the investigators will use random permuted blocks to randomize these participants into two groups. One group will have immediate Xpert test (intervention group) as the initial diagnostic test and another group will continue usual care without immediate Xpert test (control group).

Group A (Immediate NAA by clinician): NAA as the initial diagnostic test for pulmonary TB requested by clinicians.

Group B (Immediate NAA as intervention): NAA as the initial diagnostic test for pulmonary TB not requested by clinicians, but is performed as intervention in this study (intervention group).

Group C (No immediate NAA): NAA as the initial diagnostic test for pulmonary TB not requested by clinicians, and is not performed as the initial diagnostic test in this study (control group). NAA may be ordered at a later point in time by clinicians as an add-on test after sputum smear microscopy.

The investigators will assess pulmonary TB cases detected in all groups regarding

1. The interval between sputum examinations and initiation of ant-TB treatment.
2. The proportion of culture confirmed pulmonary TB among all pulmonary TB cases notified.
3. The proportion of TB patients who are advised to stop anti-TB treatment before completion of a treatment course.
4. Outcome of tuberculosis treatment, including patients who die before anti-TB treatment.

Among patients with NAA as the initial diagnostic test (Group A and Group B), the investigators will investigate

1. Performance (sensitivity, specificity and predictive values) of NAA in the diagnosis of culture positive pulmonary TB.
2. The incremental yield of the second and third smear in patients who have both NAA test and smear microscopy as the initial diagnostic test, aiming to determine the contribution of the second and third smear in the diagnosis of pulmonary TB.
3. The proportion of NAA positive cases who were culture negative.

ELIGIBILITY:
Inclusion Criteria:

* All presumptive tuberculosis cases who have sputum examinations for the diagnosis of pulmonary TB

Exclusion Criteria:

* Tuberculosis cases who have been on treatment for 14 or more days who have sputum examinations for follow-up

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6900 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic turnaround time | through study completion, an average of 1 year
  The interval between sputum examinations and initiation of ant-TB treatment

SECONDARY OUTCOMES:
culture positive pulmonary TB | through study completion, an average of 1 year
  The proportion of culture confirmed pulmonary TB among pulmonary TB cases notified
change diagnosis | 12 months after the initiation of anti-tuberculosis treatment
  The proportion of TB patients who are advised to stop anti-TB treatment before completion of a treatment course
treatment outcomes | 12 months after the initiation of anti-tuberculosis treatment
  The proportion of patients who die before anti-TB treatment, who are successfully treated, who died during treatment, who are loss-to-follow-up, who have treatment failure and who are transferred out

OTHER OUTCOMES:
performance of nucleic acid amplification test | through study completion, an average of 1 year
  sensitivity, specificity and predictive values of nucleic acid amplification test in the diagnosis of culture positive pulmonary TB
incremental yield | through study completion, an average of 1 year
  The incremental yield of the second and third smear in patients who have both NAA test and smear microscopy as the initial diagnostic test, aiming to determine the contribution of the second and third smear in the diagnosis of pulmonary TB
NAA false positive | through study completion, an average of 1 year
  The proportion of nucleic acid amplification test positive cases who were culture negative

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Yuan Chiang, MD,DrPhilos, Principal Investigator — Wan Fang Hospital, Taipei Medical University, Taiwan
Locations (5):
- Taiwan (5):
  - Chang-Hua Hospital, Chang-hua
  - Buddhist Tzu Chi General Hospital, Hualien City
  - Taichung Veterans General Hospital, Taichung
  - Chest Hospital, Ministry of Health and Welfare, Tainan
  - Wan Fang Hospital, Taipei Medical University, Taipei

IPD SHARING:
Plan to Share IPD: Yes
individual participant data will be available on request for researchers who meet the criteria for access to confidential data
Supporting Information: Study Protocol
Time Frame: 1 year after publication of findings
Access Criteria: researchers who have been trained for research, are interested in diagnostic turnaround time of pulmonary TB, and will not use the data for commercial or publication purpose.

REFERENCES:
- [Result] Chiang CY, Enarson DA, Bai KJ, Suo J, Wu YC, Lin TP, Luh KT. Factors associated with a clinician's decision to stop anti-tuberculosis treatment before completion. Int J Tuberc Lung Dis. 2008 Apr;12(4):441-6. PMID 18371272
- [Result] Chiang CY, Chang CT, Chang RE, Li CT, Huang RM. Patient and health system delays in the diagnosis and treatment of tuberculosis in Southern Taiwan. Int J Tuberc Lung Dis. 2005 Sep;9(9):1006-12. PMID 16158893
- [Result] Chen CC, Chiang CY, Pan SC, Wang JY, Lin HH. Health system delay among patients with tuberculosis in Taiwan: 2003-2010. BMC Infect Dis. 2015 Nov 2;15:491. doi: 10.1186/s12879-015-1228-x. PMID 26527404
- [Result] Pan SC, Chen YC, Wang JY, Sheng WH, Lin HH, Fang CT, Chang SC. Tuberculosis in Healthcare Workers: A Matched Cohort Study in Taiwan. PLoS One. 2015 Dec 17;10(12):e0145047. doi: 10.1371/journal.pone.0145047. eCollection 2015. PMID 26679188
- [Result] Boehme CC, Nicol MP, Nabeta P, Michael JS, Gotuzzo E, Tahirli R, Gler MT, Blakemore R, Worodria W, Gray C, Huang L, Caceres T, Mehdiyev R, Raymond L, Whitelaw A, Sagadevan K, Alexander H, Albert H, Cobelens F, Cox H, Alland D, Perkins MD. Feasibility, diagnostic accuracy, and effectiveness of decentralised use of the Xpert MTB/RIF test for diagnosis of tuberculosis and multidrug resistance: a multicentre implementation study. Lancet. 2011 Apr 30;377(9776):1495-505. doi: 10.1016/S0140-6736(11)60438-8. Epub 2011 Apr 18. PMID 21507477
- [Result] Hermans S, Caldwell J, Kaplan R, Cobelens F, Wood R. The impact of the roll-out of rapid molecular diagnostic testing for tuberculosis on empirical treatment in Cape Town, South Africa. Bull World Health Organ. 2017 Aug 1;95(8):554-563. doi: 10.2471/BLT.16.185314. Epub 2017 Apr 28. PMID 28804167
- [Result] Cox H, Dickson-Hall L, Ndjeka N, Van't Hoog A, Grant A, Cobelens F, Stevens W, Nicol M. Delays and loss to follow-up before treatment of drug-resistant tuberculosis following implementation of Xpert MTB/RIF in South Africa: A retrospective cohort study. PLoS Med. 2017 Feb 21;14(2):e1002238. doi: 10.1371/journal.pmed.1002238. eCollection 2017 Feb. PMID 28222095
- [Result] Cox HS, Mbhele S, Mohess N, Whitelaw A, Muller O, Zemanay W, Little F, Azevedo V, Simpson J, Boehme CC, Nicol MP. Impact of Xpert MTB/RIF for TB diagnosis in a primary care clinic with high TB and HIV prevalence in South Africa: a pragmatic randomised trial. PLoS Med. 2014 Nov 25;11(11):e1001760. doi: 10.1371/journal.pmed.1001760. eCollection 2014 Nov. PMID 25423041
- [Result] Naidoo P, Dunbar R, Lombard C, du Toit E, Caldwell J, Detjen A, Squire SB, Enarson DA, Beyers N. Comparing Tuberculosis Diagnostic Yield in Smear/Culture and Xpert(R) MTB/RIF-Based Algorithms Using a Non-Randomised Stepped-Wedge Design. PLoS One. 2016 Mar 1;11(3):e0150487. doi: 10.1371/journal.pone.0150487. eCollection 2016. PMID 26930400
- [Result] Calligaro GL, Zijenah LS, Peter JG, Theron G, Buser V, McNerney R, Bara W, Bandason T, Govender U, Tomasicchio M, Smith L, Mayosi BM, Dheda K. Effect of new tuberculosis diagnostic technologies on community-based intensified case finding: a multicentre randomised controlled trial. Lancet Infect Dis. 2017 Apr;17(4):441-450. doi: 10.1016/S1473-3099(16)30384-X. Epub 2017 Jan 5. PMID 28063795
- [Result] Mbonze NB, Tabala M, Wenzi LK, Bakoko B, Brouwer M, Creswell J, Van Rie A, Behets F, Yotebieng M. Xpert((R)) MTB/RIF for smear-negative presumptive TB: impact on case notification in DR Congo. Int J Tuberc Lung Dis. 2016 Feb;20(2):240-6. doi: 10.5588/ijtld.15.0177. PMID 26792478
- [Result] Automated Real-Time Nucleic Acid Amplification Technology for Rapid and Simultaneous Detection of Tuberculosis and Rifampicin Resistance: Xpert MTB/RIF Assay for the Diagnosis of Pulmonary and Extrapulmonary TB in Adults and Children: Policy Update. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK258608/ PMID 25473701
- [Result] Lin HH, Dowdy D, Dye C, Murray M, Cohen T. The impact of new tuberculosis diagnostics on transmission: why context matters. Bull World Health Organ. 2012 Oct 1;90(10):739-747A. doi: 10.2471/BLT.11.101436. Epub 2012 Jul 16. PMID 23109741
- [Result] Steingart KR, Schiller I, Horne DJ, Pai M, Boehme CC, Dendukuri N. Xpert(R) MTB/RIF assay for pulmonary tuberculosis and rifampicin resistance in adults. Cochrane Database Syst Rev. 2014 Jan 21;2014(1):CD009593. doi: 10.1002/14651858.CD009593.pub3. PMID 24448973
- [Result] Mase SR, Ramsay A, Ng V, Henry M, Hopewell PC, Cunningham J, Urbanczik R, Perkins MD, Aziz MA, Pai M. Yield of serial sputum specimen examinations in the diagnosis of pulmonary tuberculosis: a systematic review. Int J Tuberc Lung Dis. 2007 May;11(5):485-95. PMID 17439669
- [Result] Lombardi G, Di Gregori V, Girometti N, Tadolini M, Bisognin F, Dal Monte P. Diagnosis of smear-negative tuberculosis is greatly improved by Xpert MTB/RIF. PLoS One. 2017 Apr 21;12(4):e0176186. doi: 10.1371/journal.pone.0176186. eCollection 2017. PMID 28430807
- [Result] Ford I, Norrie J. Pragmatic Trials. N Engl J Med. 2016 Aug 4;375(5):454-63. doi: 10.1056/NEJMra1510059. No abstract available. PMID 27518663
- [Result] Rieder HL, Chiang CY, Rusen ID. A method to determine the utility of the third diagnostic and the second follow-up sputum smear examinations to diagnose tuberculosis cases and failures. Int J Tuberc Lung Dis. 2005 Apr;9(4):384-91. PMID 15830743